CLINICAL TRIAL: NCT03979417
Title: Identification of Biomarkers Related to Liver Fibrosis as New Therapeutic Targets
Acronym: FIBROTHER
Status: Completed | Type: Observational
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-069
Record Dates: First submitted 2019-04-10; First posted 2019-06-07 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-03

CONDITIONS: Hepatopathy; Fibrosis
Keywords: Biomarkers
MeSH Terms: conditions — Digestive System Diseases; Fibrosis | interventions — Blood Specimen Collection; Hepatectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood Mononuclear Cell (PBMC), Liver samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Liver fibrosis F0-F1: Blood draw and liver resection at the liver surgery
  Interventions: Other: Blood draw and liver resection
- Liver fibrosis F2-F3: Blood draw and liver resection at the liver surgery
  Interventions: Other: Blood draw and liver resection
- Liver Fibrosis F4: Blood draw and liver resection at the liver surgery
  Interventions: Other: Blood draw and liver resection

INTERVENTIONS:
Other: Blood draw and liver resection — The samples are transferred to the research unit for immunological studies.

SUMMARY:
Fibrosis is a dynamic process resulting from the balance of fibrogenesis and fibrolysis, mainly secondary to chronic necro-inflammation related to regular alcohol consumption, metabolic syndrome (NASH) or viral hepatitis. The liver has the property of allowing the reversion of fibrosis / cirrhosis when the necrotic-inflammatory activity is controlled. The balance between fibrosis / fibrolysis and its inhibition depends on many pathways and the hypothesis of the efficacy of a single treatment remains uncertain. Molecular factors in the progression of liver fibrosis should be determined. It is necessary to control the liver fibrosis and thus reduce the risk of carcinoma in this population. The anti-fibrotic drugs are being developed, but so far only alpha-tocopherol and obeticholic acid have been shown to have a significant anti-fibrotic effect in humans. Several new drugs are currently being evaluated in ongoing Phase 2 and 3 randomized clinical trials, but most of them have intrinsic limitations: (i) they take a long time for evaluation (> 3 years), ( ii) they generally require an histopathological evaluation by serial liver biopsies that are invasive and unpopular with patients who are aware of noninvasive tests for fibrosis assessment and (iii) treatment is often a single treatment versus a placebo group with the uncertainty that at 1 or 3 years, serial liver biopsies results are convincing.

DETAILED DESCRIPTION:
The study will be performed in 30 patients. Patients will be enrolled in two investigators sites (Cochin Hospital, Pitie-Salpetriere Hospital, France) where the patient selection will be conducted during a Multidisciplinary Collaborative Meeting.

The patients will be enrolled after collecting their informed consent. As soon as the patient is included, arrangements will be made for the organization of the liver resection according to the usual procedure of the hospital department.

The biological samples for the research (blood and liver) will be taken at the time of the surgery and sent to the Research Unit (Institut Pasteur) where immunological analyses will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years
* Patients with primary liver disease or liver metastases
* Patients undergoing liver resection

Exclusion Criteria:

* Presence of Human Immunodeficiency Virus (HIV) infection
* Presence of Human T Leukemia Virus (HTLV) infection
* Taking immunosuppressive drugs in the 6 months prior to surgery
* A person deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary hepatopathies or liver metastasis with indication for liver resection.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Identification of biomarkers of liver fibrosis | Baseline
  Frequency of cell receptors (CD4, CD8, NK, MAIT, etc.) in whole blood and liver (measured by FACS). A comparison will be made in each of the 3 groups (F0-F1, F2-F3, F4) and between the three groups.

SECONDARY OUTCOMES:
Transcription factors | Baseline
  Frequency of transcription factors (Stat1, Stat3, Foxp3, etc.) in whole blood and liver (measured by FACS). A comparison will be made in each of the 3 groups (F0-F1, F2-F3, F4) and between the three groups.
Evaluation of anti-fibrotic properties of biomarkers | Baseline
  Monitoring the properties by different techniques (ELISA, Nanostring, Immunoblotting). A comparison will be made in each of the 3 groups (F0-F1, F2-F3, F4) and between the three groups.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Pitie-Salpetriere Hospital, Paris
  - Cochin Hospital, Paris

IPD SHARING:
Plan to Share IPD: No